CLINICAL TRIAL: NCT06049160
Title: A Comparative Study Between Preoperative and Postoperative Rectal Misoprostol in the Reduction of Blood Loss During and After Elective Cesarean Section : A Double Blinded Randomized Controlled Trial
Brief Title: Comparative Study Between Preoperative and Postoperative Rectal Misoprostol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Martina Asaad
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2023-10

CONDITIONS: Blood Loss, Surgical; Blood Loss, Postoperative
Keywords: blood loss; Cesarean Section; Oxytocin; Rectal Misoprostol
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage; Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-operative and post-operative rectal misoprostol (Active Comparator): 64 participants who will receive combined pre-operative and post-operative rectal misoprostol (400μg rectal misoprostol during urinary catheter insertion just after spinal anesthesia plus 200μg after abdominal closure).
  Interventions: Drug: Misoprostol
- Post-operative rectal misoprostol (Active Comparator): 64 participants who will receive rectal misoprostol post-operative only (600μg of rectal misoprostol after closure of the Cesarean Wound)).
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — All participants will be assigned for giving misoprostol rectally either preoperative or postoperative
  Other Names: Syntocinon

SUMMARY:
Cesarean delivery (CD) is the most common major surgical procedure undergone by women around the world. Over the past two decades, there has been a witnessed increase in rates of caesarean deliveries, which continues to rise, achieving 30% in resource-rich countries and exceeding 60% in resource-limited countries. According to a Lancet report 2014, Egypt is one of the countries with the highest rates of caesarean delivery, in which the rate had reached 55.5%. The rate is almost double to three times the ideal rate of 10%-15%

DETAILED DESCRIPTION:
In resource-limited countries, postpartum hemorrhage (PPH) remains the leading cause of maternal mortality. The increased rates of caesarean delivery have been incriminated as the primary cause behind the rise in PPH. PPH after a caesarean delivery has been defined as blood loss over 1000 ml. The estimated prevalence rate of PPH is in the range of 0.6%-6.4%.

Increased blood loss after CD reflects several factors, including surgical incisions, lack of background uterine contraction, and manual removal of placenta rather than waiting for its spontaneous separation after placental bed retraction. Minimizing blood loss during delivery is an important preventive health objective aimed at reducing postpartum anemia and related morbidity .

It has been reported that the prevalence of postpartum anemia in low-income countries is approximately 50%-80%. The major cause of postpartum anemia is blood loss at delivery, especially in presence of prepartum anemia. Postpartum anemia constitutes an appreciable health problem among women of reproductive age and is associated with reduced quality of life, impaired cognition, emotional instability, and depression.

Oxytocin is routinely used by obstetricians to prevent excessive blood loss during CD. Oxytocin is the uterotonic of choice in obstetric medicine. Both the Royal College of Obstetricians and Gynecologists and the American College of Obstetricians and Gynecologists currently recommend the routine use of oxytocin (5 IU bolus dose or infusion, respectively) after the delivery of the infant as a prophylactic measure against PPH. However, oxytociin is a dangerous drug with serious adverse effects such as hypotension, tachyc ardiaand myocardial ischemia .

Misoprostol is a prostaglandin E1 analogue that effectively prevents and treats PPH owin g to its uterotonic properties. It can be used through different routes: oral; sublingual; bucc al; rectal; and intrauterine with similar efficacy to oxytocin in reducing blood loss. The benefits of misoprostol (cervical dilation and uterine contractions) and its adverse effects (nausea, vomiting, diarrhea, fever, and chills) are dose dependent .

Misoprostol is affordable and widely available, easily administered via multiple routes ( vaginal, rectal, sublingual, and oral), and has a good safety profile if properly administered and monitored, all of which make it the standard treatment option for PPH in low-resource settings.

Misoprostol administered vaginally is affected by vaginal acidity and the bacterial micro-environment. Sublingual route has the highest peak concentration; however, it is also associated with the highest incidence of adverse effects due to high peak concentrati on. Rectally administered misoprostol is associated with slower absorption, lower peak c oncentration levels, and reduced adverse effects compared with the oral and sublingua l routes.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age ( 37 to 41 weeks).
2. Singleton healthy fetus.
3. Scheduled for elective lower segment caesarean delivery under spinal anaesthesia.
4. Body mass index of (25-30 Kg/m2).
5. Normal coagulation profile.
6. Normal amniotic fluid volume assessed by amniotic fluid index.

Exclusion Criteria:

1. Maternal comorbidity: Hypertension; diabetes; heart, kidney, or liver disorders.
2. Contraindication to use of misoprostol like known allergy to misoprostol or asthmatic patients.
3. Women who had undergone any previous uterine surgery such as myomectomy because it is considered upper uterine segment operation with more destruction in myometrium but caesarean section is a lower segment uterine operation with minimal destruction in myometrium.
4. Women at higher risk of intraoperative blood loss or PPH, such as those with hemoglobin levels less than 9 g/dl, history of PPH, or uterine fibroids.
5. Antepartum hemorrhage ( placenta previa and placental abruption).
6. Women who will undergo caesarean section because of failure of induction of labor.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss (defined as blood loss ≥500 cc) | First 2 hours from the starting of the operation
  Outcome of the study will be measured in terms of assessment of Hemoglobin level
Intraoperative blood loss (defined as blood loss ≥500 cc) | First 2 hours from the starting of the operation
  Outcome of the study will be measured in terms of assessment of Hematocrit level

SECONDARY OUTCOMES:
Occurrence of primary postpartum hemorrhage ( defined as excessive blood loss as 1000cc during first 24 hours) | first 24 hours after C-Section]
  Outcome of the study will be measured in terms of assessment of Hemoglobin level post operatively.
Occurrence of primary postpartum hemorrhage ( defined as excessive blood loss as 1000cc during first 24 hours) | first 24 hours after C-Section]
  Outcome of the study will be measured in terms of assessment of Hematocrit level post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Khayat, Professor, Study Chair — Cairo University
Locations (1):
- Faculty of medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided